CLINICAL TRIAL: NCT04925908
Title: Evaluation of Exclusive Breastfeeding Within the First Six Months in Infants of Mothers Infected With Novel Coronavirus: 1-year Experience of a Single Center
Brief Title: Exclusive Breastfeeding in Infants of Mothers Infected With Novel Coronavirus
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.05.165
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Covid19; Breastfeeding, Exclusive; Newborn Morbidity
MeSH Terms: conditions — COVID-19; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Infants of mothers with suspected but negative for COVID-19
  Interventions: Diagnostic Test: RT-PCR for SARS-Cov-2
- Case Group: Infants Born to COVID-19 positive mothers
  Interventions: Diagnostic Test: RT-PCR for SARS-Cov-2

INTERVENTIONS:
Diagnostic Test: RT-PCR for SARS-Cov-2 — Nasopharyngeal swab for detecting Novel Coronavirus-2 by reverse transcriptase polymerase chain reaction

SUMMARY:
COVID-19 pandemic emerges an issue for breastfeeding.Earlier in pandemic mothers who had COVID-19 were separated from their babies due to insufficient data but this approach was abandoned due to the lack of transmission via breastmilk.However, where mothers with COVID-19 are cohorted in the same room, they still have to be isolated from their babies following the birth.Investigators aimed to evaluate rate of exclusive breastfeeding(EB) within first 6 months among mothers who were isolated from their babies due to COVID-19.

DETAILED DESCRIPTION:
COVID-19 pandemic emerges an issue for breastfeeding.Earlier in pandemic mothers who had COVID-19 were separated from their babies due to insufficient data but this approach was abandoned due to the lack of transmission via breastmilk.However, where mothers with COVID-19 are cohorted in the same room, they still have to be isolated from their babies following the birth.To our knowledge, there is no study regarding this subject to-date.Therefore, investigators aimed to evaluate rate of exclusive breastfeeding(EB) within first 6 months among mothers who were isolated from their babies due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Infants who were born to mothers with suspected or evident COVID-19
* Accepted to participate with an informed consent of parents

Exclusion Criteria:

* Congenital abnormalities
* Chromosomal abnormalities
* Contraindication for breastfeeding
* Declined to participate

Max Age: 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who were born to mothers with suspected/proven COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding | 6 months
  Rate of exclusive breastfeeding

SECONDARY OUTCOMES:
Disease status | 6 months
  COVID-19 positive/negative

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.